CLINICAL TRIAL: NCT02424422
Title: The Effect of Rapid Maxillary Expansion on Craniofacial Sutures in Children Using Cone Beam Computed Tomography
Brief Title: The Effect of Expansion on Craniofacial Sutures in Children Using 3D Imaging
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDDS-Ortho-01-2015
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Skeletal Maxillary Transverse Deficiency
Keywords: Corrective Orthodontics; CBCT; Rapid Maxillary Expansion; Cone Beam Computed Tomography; Hyrax Expansion; Craniofacial Sutures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study to test the immediate effect of rapid maxillary expansion on craniofacial sutures in children using cone beam computed tomography.

Materials and Methods: Subjects consisted of 15 growing patients between the ages of 8 and 12 with Skeletal transverse maxillary deficiency with unilateral or bilateral posterior cross bite.

All patients will be treated with A bonded Hyrax (a rapid palatal expander with an acrylic occlusal splint). The planned activation protocol consisted of 2 turns per day (0.25 mm per turn) until the resolution of posterior cross bite with 2 to 3 mm overcorrection of expansion then tying off the jackscrew with a ligature wire and placing a smooth composite material over it. The initial CBCT scan (T0) will be taken before cementation of the maxillary expander and again immediately after the end of the active expansion (T1). First, all CBCT images will be oriented then the craniofacial sutures(Intermaxillary Suture, Midpalatal Suture, Transpalatal Suture, Internasal Suture, Frontonasal suture, Zygomaticotemporal suture, Frontomaxillary suture, Zygomaticomaxillary suture, Nasomaxillary sutures, Spheno-occipital synchondrosis) will be examined. Where the linear measurements will be carried out directly on the CBCT image using the OnDemand 3D Imaging software program.

DETAILED DESCRIPTION:
Rapid maxillary expansion (RME) treatment has been used widely since the mid 1960s. It is frequently used to correct maxillary width deficiency, posterior crossbite or to expand arch perimeters to alleviate dental crowding or patients with Class III malocclusion who often are treated with RME because of an insufficient maxillary arch width. Although, the major effect of this treatment is noticed clinically in the dentition and maxilla area. RME therapy appears to involve an ample portion of the craniofacial complex, as the maxilla is associated with 10 bones in the face and head. Although, the RME force is concentrated on widening the maxilla, concomitant changes occur in circumaxillary sutures. Moreover, it has been claimed that the transverse forces generated during rapid maxillary expansion are transmitted, via the pterygomaxillary connection, to the unpaired sphenoid bone of the cranial base, where they lead to stress. The extent and effects of this have not yet been studied extensively, nor have they been well determined. In orthodontics, the cranial base has received attention because of the fact that its growth influences the maxillary-mandibular complex. Some authors in fact consider the cranial base as a guide rail for development of the maxilla, midface, and lower facial complex. This involvement has been hypothesized following investigations based on histologic methods, radiologic imaging, photoelastic models, bone scintigraphy, and finite element analysis. However, even though the above studies have been well designed, some issues may have affected their conclusions. In fact, histological findings are limited to experimental studies in animals. Moreover, accuracy of the results of the finite element model (FEM) depends on the detailed geometry, material properties, and boundary conditions of the FEM. Therefore, until now, there have been only speculations about whether RME can or cannot disarticulate these structures in humans. With advanced technology and the introduction of three-dimensional computed tomography imaging, that allow clinicians and researchers to quantitatively evaluate bone changes with minimal distortion and lower radiation dosage, Due to the high dose of x-ray of CT, high cost and the lack of study on the effect of the RME on circumaxillary sutures and spheno-occipital synchondrosis using imaging three-dimensional radiographic (CT). Because of the importance of the effect of the maxillary expansion on maxillary displacement, and the resulting significant clinical effects, especially at the level of improvement in the third class at the children. From here stems the need for this study on the effect of rapid maxillary expansion RME on the craniofacial sutures in children using cone beam computed tomography

ELIGIBILITY:
Inclusion Criteria:

* skeletal maxillary transverse deficiency
* age between 8 and 12
* not previously treated orthodontically
* no presence of craniofacial syndromes or congenital deformities
* presence of unilateral or bilateral cross-bites

Exclusion Criteria:

* previous orthodontic treatment
* absence of any posterior cross-bite
* presence of any congenital malformations or dentofacial syndromes
* patients of non-Syrian ancestry
* mental retardation

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Growing patients between the age of 8 and 12 will be recruited from those who are visiting the Department of Orthodontics at University of Damascus Dental School.
  The study will evaluate the impact of maxillary expansion on craniofacial sutures using CBCT imaging.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in craniofacial suture width | A CBCT image will be taken before the commencement of maxillary expansion and anther CBCT image will be taken within 3 days following orthopedic appliance removal
  The distance between the two edges of each suture.
  The following sutures will be measured:
  Intermaxillary Suture, Midpalatal Suture, Transpalatal Suture, Internasal Suture, Frontonasal suture, Zygomaticotemporal suture, Frontomaxillary suture, Zygomaticomaxillary suture, Nasomaxillary sutures, Spheno-occipital synchondrosis

CONTACTS AND LOCATIONS:
Overall Officials: Nemat Al-Kaissi, DDS, Principal Investigator — MSc student at the Department of Orthodontics, University of Damascus Dental School; Mowaffak Ajaj, DDS MSc PhD, Study Director — Associate Professor of Orthodontics, University of Damascus Dental School
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Damascsus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bazargani F, Feldmann I, Bondemark L. Three-dimensional analysis of effects of rapid maxillary expansion on facial sutures and bones. Angle Orthod. 2013 Nov;83(6):1074-82. doi: 10.2319/020413-103.1. Epub 2013 Jun 7. PMID 23745976
- [Background] Leonardi R, Cutrera A, Barbato E. Rapid maxillary expansion affects the spheno-occipital synchondrosis in youngsters. A study with low-dose computed tomography. Angle Orthod. 2010 Jan;80(1):106-10. doi: 10.2319/012709-56.1. PMID 19852648
- [Background] Leonardi R, Sicurezza E, Cutrera A, Barbato E. Early post-treatment changes of circumaxillary sutures in young patients treated with rapid maxillary expansion. Angle Orthod. 2011 Jan;81(1):36-41. doi: 10.2319/050910-250.1. PMID 20936952
- [Background] Gardner GE, Kronman JH. Cranioskeletal displacements caused by rapid palatal expansion in the rhesus monkey. Am J Orthod. 1971 Feb;59(2):146-55. doi: 10.1016/0002-9416(71)90046-7. No abstract available. PMID 4993115
- [Background] Lee H, Ting K, Nelson M, Sun N, Sung SJ. Maxillary expansion in customized finite element method models. Am J Orthod Dentofacial Orthop. 2009 Sep;136(3):367-74. doi: 10.1016/j.ajodo.2008.08.023. PMID 19732671
- [Background] Mah JK, Huang JC, Choo H. Practical applications of cone-beam computed tomography in orthodontics. J Am Dent Assoc. 2010 Oct;141 Suppl 3:7S-13S. doi: 10.14219/jada.archive.2010.0361. PMID 20884934